CLINICAL TRIAL: NCT02178943
Title: Utility of Donor-Derived Cell-free DNA in Association With Gene-Expression Profiling (AlloMap®) in Heart Transplant Recipients (D-OAR)
Brief Title: Utility of Donor-Derived Cell Free DNA in Association With Gene Expression Profiling
Acronym: D-OAR
Status: Completed | Type: Observational
Sponsor: CareDx (Industry)
Responsible Party: Sponsor
Other Study IDs: SN-C-00004
Record Dates: First submitted 2014-06-13; First posted 2014-07-01 (Estimated); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Cardiac Transplant Failure; Cardiac Transplant Rejection; Heart Diseases
Keywords: Molecular Diagnostics; Heart Transplantation; Risk Factors; Prognosis
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — donor derived cf-DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart Transplant Recipients: Heart allograft recipients undergoing scheduled surveillance visits that are part of a long-term management plan.

SUMMARY:
Plasma donor-derived cell-free DNA (dd-cfDNA) is measured as a % of the total plasma cfDNA in association with the measurement of AlloMap, a non-invasive gene expression test to aid in heart transplant management.

DETAILED DESCRIPTION:
AlloMap Molecular Expression Testing is performed in a single laboratory, assessing the gene expression profile of RNA isolated from peripheral blood mononuclear cells (PBMC). Per FDA labeling, AlloMap Testing is "intended to aid in the identification of heart transplant recipients with stable allograft function who have a low probability of moderate/severe acute cellular rejection (ACR) at the time of testing in conjunction with standard clinical assessment." AlloMap is the only non-invasive, blood test method recommended in the International Society for Heart and Lung Transplantation (ISHLT) guidelines for surveillance of heart transplant recipients for rejection. More than 52,000 commercial AlloMap tests from more than 12,000 patients have been reported by the XDx Reference Laboratory in Brisbane, California, which is certified under the Clinical Laboratory Improvement Amendment (CLIA) of 1988 and accredited by the College of American Pathologists.

In 2013, a registry study named OAR was initiated to follow long-term outcomes in allograft recipients receiving commercial AlloMap testing for surveillance (NCT01833195). The current objective is to enroll volunteers who are participating in the OAR registry(1) to co-participate in this observational sub-study, named D-OAR, in order to study a new biomarker, dd-cfDNA.

dd-cfDNA has been proposed as a marker for cellular injury caused by rejection(2, 3). Because dd-cfDNA and the AlloMap test measure different signals in the blood, a combination of the two approaches could be additive since AlloMap is a measure of host immune response and dd-cfDNA monitors graft injury.

The dd-cfDNA measurement is intended for the quantitative detection of plasma dd-cfDNA as a % of the total plasma cell-free DNA. Its utility as a surveillance tool in the management of heart transplant recipients is being investigated.

This is an observational sub-study for subjects who are co-enrolled to participate in the Outcomes AlloMap Registry (OAR). Prior to implementation of the amendment dated September 15, 2016, blood specimens were collected for assay of dd-cfDNA levels at each visit that occurred for AlloMap testing, per the OAR Study. As stated in the OAR study, the regular surveillance schedule for testing with AlloMap is determined by each participating center's standard of care. After this protocol amendment, the existing patients will no longer have routine dd-cfDNA specimens drawn to be paired with their standard of care AlloMap. The dd-cfDNA specimen will be drawn only when the patient is scheduled for a for-cause biopsy. New patients may be enrolled any time post-transplant as long as they have not had more than 1 prior AlloMap. These patients will also only undergo routine AlloMap testing as per participating center's standard of care and dd-cfDNA specimen will be drawn when the patient is scheduled for a for-cause biopsy. An AlloMap sample will be drawn for research use along with the dd-cfDNA specimen at the time of the for-cause biopsy where the center's infrastructure permits. An additional two follow-up dd-cfDNA specimens will be collected in the patients that undergo a for-cause biopsy, and are being treated for rejection and/or graft dysfunction, as per their standard of care schedule. The two follow-up visits will not be paired with a research use AlloMap and will be performed within 8 weeks after the for cause event. If a patient returns for another for-cause biopsy, the center may opt to collect another research AlloMap and dd-cfDNA specimen, and two follow-up dd-cfDNA specimens.

ELIGIBILITY:
Inclusion Criteria

1. Any heart transplant recipient eligible for initiation and participation in the Outcomes AlloMap Registry (OAR) Study of regular AlloMap testing.
2. Patients can be enrolled any time as long as they have not had more than 1 prior AlloMap.
3. Written informed consent must be obtained prior to study enrollment. Exclusion Criteria

1. Pregnant Women.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Heart allograft recipients undergoing scheduled surveillance visits that are part of a long-term management plan.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-06; Primary Completion 2019-12 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Clinical Outcomes (Vital Status of Heart Transplant Recipients) | 3 years
  Graft dysfunction, Rejection with hemodynamic compromise:
  Hemodynamic compromise is defined by the presence of one or more of the following criteria:
  Proportional decrease in LVEF ≥ 25%, Absolute LVEF ≤ 30%, Need for inotropic support, Cardiac index < 2.0 L/min/m2, Death (re-transplantation)

CONTACTS AND LOCATIONS:
Overall Officials: James P Yee, Study Director — CareDx Inc (formerly XDx Inc) Brisbane, CA
Locations (28):
- United States (28):
  - Cedars-Sinai Medical Center, Beverly Hills, California
  - University of California, Los Angeles, Los Angeles, California
  - Stanford University, Stanford, California
  - Memorial Regional Hospital, Hollywood, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - St. Vincent Medical Group, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mid America Heart Institute - St. Luke's Hospital, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - Columbia University Medical Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Drexel University, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor Research Institute, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor St. Lukes, Houston, Texas
  - Intermountain Heart Institute, Murray, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Background] Grskovic M, Hiller DJ, Eubank LA, Sninsky JJ, Christopherson C, Collins JP, Thompson K, Song M, Wang YS, Ross D, Nelles MJ, Yee JP, Wilber JC, Crespo-Leiro MG, Scott SL, Woodward RN. Validation of a Clinical-Grade Assay to Measure Donor-Derived Cell-Free DNA in Solid Organ Transplant Recipients. J Mol Diagn. 2016 Nov;18(6):890-902. doi: 10.1016/j.jmoldx.2016.07.003. Epub 2016 Oct 7. PMID 27727019
- [Result] Kobashigawa, JA. et al; Initial Analysis of the Donor-Derived Cell-Free DNA -Outcomes AlloMap Registry (D-OAR) Study in Heart Transplant Recipients Undergoing Surveillance for Rejection. 2016 ISHLT 36th Annual Meeting and Scientific Sessions. April 27-30, 2016; Washington, DC